CLINICAL TRIAL: NCT00148460
Title: A Randomised, Open-label, Multi-center, Angiographic Trial to Compare the Efficacy and Safety of Single Bolus of Tenecteplase (Metalyse®) With Accelerated Infusion of Alteplase in Asian Patients With Acute Myocardial Infarction
Brief Title: Trial to Compare the Efficacy and Safety of a Single Bolus of TNK-tPA (Tenecteplase, Metalyse®) With Accelerated Infusion of Rt-PA (Alteplase, Actilyse®) in Asian Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.8
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — TNK-tissue plasminogen activator

INTERVENTIONS:
Drug: TNK-tPA
Drug: rt-PA

SUMMARY:
The objective of this trial was to compare the efficacy and safety of a single bolus of TNK-tPA (tenecteplase, Metalyse®) compared with rt-PA (alteplase, Actilyse®) in Asian patients.

DETAILED DESCRIPTION:
This was a randomized (1:1), open-label, multi-center, active-control, parallel-group study to compare the efficacy and safety of TNK-tPA (tenecteplase, Metalyse®) with that of accelerated rt-PA (alteplase, Actilyse®) in Asian patients with AMI. The primary endpoint (TIMI 3 Flow) and the secondary endpoint (TIMI frame count) were evaluated in a blinded manner in the core laboratory.

Patients eligible for the trial who met all inclusion and exclusion criteria and who gave their informed consent were randomized to one of two treatment groups (i.e. TNK-tPA or accelerated rt-PA).

The study period totaled 30-37 days and included baseline, randomisation, study drug administration, in-hospital follow-up and thirty-day follow-up.

Coronary angiography was performed at 90 minutes after the start of study drug administration. 12-lead electrocardiograms (ECGs) were obtained before randomization, between 60 to 75 minutes and 180 ± 15 minutes after the start of study drug administration, and at hospital discharge.

If the patient showed rapid and progressive hemodynamic deterioration before 90 minutes, rescue PTCA or other appropriate interventions should be performed at the discretion of the treating physician.

Following the analysis of TIMI flow and frame count at each study center, the results were carefully recorded on the CRFs. This data was stored on a compact disk or a film and labeled with the subject's study I.D. number. It was then sent with the summary worksheets and ECGs to the Angiographic Core Laboratory located at the Leuven Coordinating Center (LCC) of the University Hospital Gasthuisberg (Leuven, Belgium) for central evaluations.

Study Hypothesis:

The null hypothesis tested was that there was no difference between the two treatment groups: TNK-tPA (Tenecteplase, Metalyse®) and accelerated rt-PA (Actilyse®), against the alternative that there was a difference.

Comparison(s):

The primary endpoint of the study was TIMI 3 flow at 90 minutes after start of thrombolytic therapy, angiograms were evaluated in a blinded manner in a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 and <= 75 years.
2. Asian origin.
3. Ischemic discomfort >= 30 minutes in duration.
4. Onset of acute myocardial infarction (AMI) symptoms within 6 hours prior to randomization.
5. A twelve lead electrocardiogram (ECG) with one of the following:

   * ST segment elevation >= 0.1 mV in two or more limb leads; or
   * >= 0.2 mV in two or more contiguous precordial leads indicative of AMI.
6. Ability to give informed consent.

Exclusion Criteria:

1. Previous coronary artery bypass grafting (CABG) surgery.
2. Cardiogenic shock (e.g. systolic blood pressure [SBP] < 90 mmHg).
3. Systolic blood pressure (SBP) >= 180 mmHg and/or diastolic blood pressure (DBP) >= 110 mmHg during current admission on one reliable measurement prior to randomization.
4. Inability to undergo cardiac catheterization.
5. Significant bleeding disorder either at present or within the past 6 months.
6. Major surgery, biopsy of a parenchymal organ, or significant trauma within 3 months.
7. Any minor head trauma and/or any other trauma that occurred after onset of current myocardial infarction.
8. Use of heparin, GPIIb/IIIa antagonists or other anticoagulants within the last 2 weeks.
9. Any known history of stroke or transient ischemic attack or central nervous system structural damage (i.e. neoplasm, aneurysm, intracranial surgery).
10. Prolonged cardiopulmonary resuscitation (> 10 minutes) within 2 weeks.
11. Pregnancy, lactation or parturition within the previous 30 days. Women of childbearing potential must have had a negative pregnancy test and must have used a medically accepted method of birth control (i.e. uterine device, surgical sterilisation, progestogens alone).
12. Previous treatment with TNK-tPA (tenecteplase).
13. Inability to follow protocol and comply with follow-up.
14. Drug abuse within the last year.
15. Participation in another clinical trial within the previous 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2001-03; Study Completion 2006-02

PRIMARY OUTCOMES:
The percentage of patients with thrombolysis in myocardial infarction (TIMI) grade 3 flow in the infarct-related artery (IRA) | at 90 minutes after the start of thrombolytic treatment

SECONDARY OUTCOMES:
Infarct-related artery patency | at 90 minutes
The percentage of subjects with ST-segment resolution | at 60 and 180 minutes
Mortality | 30-days
Safety
The effects of TNK-tPA on coagulation and fibrinogenolysis (at selected clinical sites)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (18):
- China (9):
  - Beijing An Zhen Hospital, Beijing
  - Beijing University, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Xuan Wu Hospital, Beijing
  - Bejing Tongren Hospital, Beijing
  - Center Hospital of Dalian, Dalian
  - Center Hospital of Jinan, Jinan
  - Fudan University, Shanghai
  - People's Hospital of Liaoning Province, Shenyang
- The University of Hong Kong, Cardiology Division, Hong Kong, Hong Kong
- South Korea (8):
  - Dongsan Medical Center, Jung-Ku
  - Chunnam University Hospital, Kwangju
  - Dong-A University Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Seoul Joongang Hospital, Seoul
  - A-Jou University Hospital, Suwon
  - Wonju Christian Hospital (Yonsei University Hosp), Wŏnju